CLINICAL TRIAL: NCT04168736
Title: Family Disclosure in Cascade Testing
Status: Completed | Type: Observational
Sponsor: University of Virginia (Other)
Responsible Party: Sponsor
Other Study IDs: 19149
Record Dates: First submitted 2019-07-25; First posted 2019-11-19 (Actual); Last update posted 2019-11-19 (Actual); Status verified 2019-11

CONDITIONS: Genetic Predisposition
Keywords: genetic testing; cascade; family disclosure
MeSH Terms: conditions — Genetic Predisposition to Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Feasibility and Acceptability of Genetic Counseling Materials — To determine the feasibility and acceptability of a communication aid in sharing genetic test results with family members.
  To determine the utility of a communication aid in sharing information. To determine the impact of patient focused information sheets on patient knowledge of genetic testing.

SUMMARY:
Prospective cohort study to evaluate the feasibility and acceptability of using standardized educational and communication tools to assist in communication of genetic test results to family members. A pre and post test will be administered to consented patients before and after genetic counseling .

DETAILED DESCRIPTION:
This will be a prospective cohort study to evaluate 1) the feasibility and acceptability of using standardized educational and communication tools to assist in communication of genetic test results to family members, 2) utility of the communication tool, and 3) the impact of a patient focused information sheet on the knowledge of genetic testing in women who attend the women's oncology clinic. Genetic counseling is recommended for all women with a diagnosis of ovarian cancer, most patients with pre-menopausal diagnosis of breast cancer, and in younger women with uterine or other gynecologic malignancies. Women with a diagnosis of breast or gynecologic cancer who elect to undergo genetic testing will be approached to participate in this study. If they consent, they will be provided with two information handouts (FORCE sharing worksheets) and family letter template. Participants will complete a baseline knowledge survey prior to receipt of these materials. At a second visit, they will complete the knowledge survey again. Knowledge surveys will be scored and pre and post test scores will be compared with a paired t-test. Feasibility will be assessed by tracking the number of patients approached to participate, the number who sign consents, and the number who complete the study.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* Diagnosis of breast or gynecologic cancer
* Undergoing any genetic testing at UVA for standard clinical purposes in the Women's Oncology Clinic

Exclusion Criteria:

* Not receiving treatment at UVA
* Not English literate
* Unable to provide consent
* Known pregnancy (self-reported)

Min Age: 18 Years | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Must have a diagnosis of breast or gynecologic cancers and undergoing any genetic testing at UVA for standard clinical purposes in the Women's Oncology Clinic
Study Population: It is estimated that up to 24% of ovarian cancers are hereditary in nature, with the BRCA genes accounting for 15-18% of cases. Women with BRCA mutations have an up to 65% lifetime risk of breast cancer and an increased risk of uterine serous cancer. With implications for prognosis and treatment, the NCCN and the SGO recently endorsed universal BRCA testing for all women with ovarian cancer. Genetic counseling is recommended for women with triple negative breast cancers, pre-menopausal breast cancer with certain risk factors. Additionally, these results have implications for a patient's family. In a patient with a positive BRCA mutation, first-degree relatives have 50% chance and second-degree relatives have a 25% chance of carrying the mutation.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2017-06-30 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
percentage of family members told in comparison to number of family members | 1 year
  Evaluate the feasibility and acceptability of using standardized educational and communication tools to assist in communication of genetic test results to family members

SECONDARY OUTCOMES:
percentage of participants that report using the intervention | 1 year
  Evaluate the utility of the communication tool
To compare pre- and post test scores to accesses the gaps in traditional genetic counseling education sessions | 1 year
  Evaluate the impact of a patient focused information sheet on the knowledge of genetic testing in women who attend the women's oncology clinic

CONTACTS AND LOCATIONS:
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

DOCUMENTS (1):
  • Informed Consent Form (2017-06-30): https://cdn.clinicaltrials.gov/large-docs/36/NCT04168736/ICF_000.pdf